CLINICAL TRIAL: NCT02877342
Title: Reducing the Burden of Injury in India and Australia Through Development and Piloting of Improved Systems of Care - Prehospital Notification and Structured Handover on Hospital Arrival
Brief Title: Pre-hospital Notification of Injured Patients Presenting to Trauma Centres in India
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teresa Howard (Other)
Collaborators: National Trauma Research Institute (Other); The Alfred (Other); Monash University (Other); All India Institute of Medical Sciences (Other); The George Institute for Global Health, Australia (Other); Sheth Vadilal Sarabhai General Hospital (Other); Guru Teg Bahadur Hospital (Other); Lokmanya Tilak Municipal Medical College and Hospital (Other); Centralised Accident and Trauma Services, Delhi, India (Other Government); GVK EMRI: Emergency Management and Research Institute (Other); Maharashtra Emergency Medical Services, India (Other); Nathiba Hargovandas Lakhmichand Municipal Medical College, India (Unknown); University College of Medical Sciences, India (Individual)
Responsible Party: Sponsor-Investigator, Teresa Howard, Research Manager, National Trauma Research Institute
Organization: National Trauma Research Institute (Other)
Other Study IDs: GCF020013-PHN
Record Dates: First submitted 2016-08-03; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Major Trauma
Keywords: Injury; Injuries; Triage
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-intervention: All injured patients arriving by ambulance (to the four intervention sites) and allocated to a red (1st) or yellow (2nd) priority category will be eligible for inclusion. Patients arriving without notification buy ambulance service
- Post-Intervention: All injured patients arriving by ambulance, and allocated to a red (1st) or yellow (2nd) priority category will be eligible for inclusion. Patients arriving with and without notification by the ambulance service using the pre-hospital notification application.
  Interventions: Other: Pre-hospital notification

INTERVENTIONS:
Other: Pre-hospital notification — Pre-hospital notification smartphone/tablet application in the form of an Android program that will be used by ambulance clinicians to notify emergency departments of selected hospitals of an impending arrival of a patient.
  Other Names: Soochana app
  Groups: Post-Intervention

SUMMARY:
A prospective observational study using an interrupted time-series design to evaluate the effect of pre-hospital notification on trauma patients arriving at a trauma centre by ambulance, in India

DETAILED DESCRIPTION:
This is a longitudinal prospective cohort study of injured patients being transported by ambulance to the major trauma centre study sites. In the pre-intervention phase, prospective data on patients will be collected on pre-hospital assessment, notification, in-hospital assessment, management and outcomes and recorded in a new tailored multi-hospital trauma registry. All injured patients arriving by ambulance and allocated to a red or yellow priority category will be eligible for inclusion. The intervention will be a pre-hospital notification application in the form of an Android program that will be used by ambulance clinicians to notify emergency departments of selected hospitals of an impending arrival of a patient. The application will use a simple algorithm based on trauma triage principles developed by the Australia-India Trauma System Collaboration (AITSC). The proportion of severely injured patients arriving to hospital after notification will be the primary outcome measure with a target of 70%. Secondary outcomes evaluated will be availability of a trauma cubicle, presence of a trauma team on patient arrival, time to first chest x-ray and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria: All injured patients arriving by ambulance and allocated to a red (1st) or yellow (2nd) priority category will be eligible for inclusion. Data will be collected prospectively by trained data collectors positioned in the trauma centres.

Retrospective inclusion will be continued for all screened patients presenting to any of the included hospitals with injury (including near-drowning) as the primary diagnosis and with at least one of the following criteria:

1. Admission to hospital
2. Death after triage but before admission
3. Dead on arrival

Exclusion criteria: Patients meeting screening criteria will be subsequently excluded if they meet any of the following criteria:

1. Dead at scene
2. Alive at triage but not admitted to hospital (discharged alive)
3. Isolated poisoning
4. Isolated burns
5. Single digit finger or toe amputations (unless of the thumb or great toe), only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in four major trauma centres in India. The Jai Prakash Narayan Apex Trauma Center, All India Institute of Medical Sciences (AIIMS), New Delhi admits approximately 4000 injured patients per year. Guru Tegh Bahadur (GTB) Hospital is a 1,500-bed hospital situated in the National Capital Region of Delhi, India, with a trauma census of approx. 1500 per year. The Lokmanya Tilak Municipal General (LTMG) Hospital is a Level I trauma centre, which caters to the megapolis of Mumbai and receives about 1000 injured patients per year. The Sheth Vadilal Sarabhai General (VS) Hospital caters to areas in and around Ahmedabad with an average annual admission secondary to trauma of about 1200/year.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-08 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Pre-hospital notification | 1 - 1.5 years
  Prior to arrival at emergency department. Pre-hospital notification will be the primary outcome, defined as a phone call or message to a treating hospital clinician regarding an injured patient enroute to hospital. For the purpose of this research project, a patient will satisfy primary outcome criteria if pre-hospital notification with any information has occurred. This variable will be collected and analysed as a binary variable.

SECONDARY OUTCOMES:
Trauma Call out | 1 - 1.5 years
  A trauma callout occurs in response to the notification. A trauma call-out will be recorded as a binary variable- whether one has occurred or not.
Presence of trauma team leader | 1 - 1.5 years
  Trauma leader is present when the patient enters the emergency department for treatment. The presence of a trauma team leader at the time of patient arrival will be collected as a binary variable. This is the person whose role is to co-ordinate the trauma resuscitation
Readiness of trauma bay | 1 - 1.5 years
  At least 1 trauma bay that has been allocated and empty (therefore ready to receive a patient) on arrival.
Time to first chest x-ray | 1 - 1.5 years
  Time at which the first chest x-ray commenced will be recorded.
Location of patient discharge | 1 - 1.5 years
  The location to which a patient was discharged on completion of hospital management will be recorded
In-hospital death | 1 - 1.5 years
  Patient death whilst in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Fitzgerald, MBBS, MD, Principal Investigator — National Trauma Research Institute
Locations (4):
- India (4):
  - Vadilal Sarabhai Hospital, Ahmedabad, Gujarat
  - Guru Teg Bahadur Hospital, Delhi
  - JPN Apex Trauma Centre at All India Institute of Medical Sciences, Delhi
  - Lokmanya Tilak Municipal General Hospital, Mumbai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitra B, Kumar V, O'Reilly G, Cameron P, Gupta A, Pandit AP, Soni KD, Kaushik G, Mathew J, Howard T, Fahey M, Stephenson M, Dharap S, Patel P, Thakor A, Sharma N, Walker T, Misra MC, Gruen RL, Fitzgerald MC; Australia-India Trauma System Collaboration. Prehospital notification of injured patients presenting to a trauma centre in India: a prospective cohort study. BMJ Open. 2020 Jun 21;10(6):e033236. doi: 10.1136/bmjopen-2019-033236. PMID 32565447
- [Derived] Mitra B, Mathew J, Gupta A, Cameron P, O'Reilly G, Soni KD, Kaushik G, Howard T, Fahey M, Stephenson M, Kumar V, Vyas S, Dharap S, Patel P, Thakor A, Sharma N, Walker T, Misra MC, Gruen R, Fitzgerald M; Australia-India Trauma System Collaboration. Protocol for a prospective observational study to improve prehospital notification of injured patients presenting to trauma centres in India. BMJ Open. 2017 Jul 17;7(7):e014073. doi: 10.1136/bmjopen-2016-014073. PMID 28716784